CLINICAL TRIAL: NCT02126709
Title: Phase 2 Study of the Efficacy and Safety of 3% Povidone-Iodine in Acne Therapy
Brief Title: The Efficacy and Safety of 3% Povidone-Iodine in Acne Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Mundipharma Pte Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013/01233
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Acne
Keywords: Povidone Iodine; Safety; Efficacy; Acne treatment
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm (Experimental): Name: Repigel Active ingredient: Povidone iodine Dosage form: Liposomal hydrogel Administration route: Topical Strength: 3%
  Application of study cream twice a day during the 8 week study period
  * It will be applied once in the morning and once in the night
  * We recommend the application to occur after the face is washed
  * One Finger Tip Unit is required per application to the entire face
  * The gel should be left on and not washed of for at least15 -30 minutes
  Interventions: Drug: Repigel
- Placebo Arm (Placebo Comparator): Name: Neutrogena hydroboost gel Active ingredient: NA Strength: NA Dosage form: Water gel Administration route: Topical
  Application of placebo cream twice a day during the 8 week study period
  * It will be applied once in the morning and once in the night
  * We recommend the application to occur after the face is washed
  * One Finger Tip Unit is required per application to the entire face
  * The gel should be left on and not washed of for at least15 -30 minutes

INTERVENTIONS:
Drug: Repigel — Repigel will be used as the intervention in the treatment group
  Arms: Treatment Arm

SUMMARY:
Importance This will be a proof of concept study - whereby we hypothesize that Repigel may represent a paradigm shift in global acne treatment.

Historically, there has been a dearth of clinical evidence in this use of povidone-iodine for inflammatory acne. This is likely due to staining related to iodine use, which is not acceptable to consumers.

The trial drug, Povidone Iodine, however, becomes colourless and odourless in a matter of seconds after application on the skin.

This represents an ideal product for which we may perform testing to look at its efficacy in the management of acne.

A mainstay in the pathogenesis of acne involves the overgrowth and proliferation of skin micro-organisms, primarily proprionibacterium Acnes. Long term antibiotic therapy is usually prescribed for a period of 3 to 6 months or more.

Previous studies have revealed this form of antibiotic therapy is ineffective, patients are usually poorly compliant, and also results in the formation of antibiotic resistant micro-organisms,which in turn reduces treatment efficacy.

Potential Benefits

As such, Povidone Iodine with its antiseptic property represents a promising avenue for the elimination of Proprionibacterium Acnes without the associated problems of long term antibiotic use, and the development of antibiotic-resistance. It is cosmetically acceptable, affordable, and easy to use.

DETAILED DESCRIPTION:
Aim This is a proof of concept study - to determine the efficacy and safety of Povidone Iodine in the treatment of acne.

Methodology This will be a single centre, double blind, randomized controlled trial. There will be 2 arms of 15 patients with a 2 month study period.

Follow up at Week 0, Week 2, Week 4, Week 6, Week 8

3. Capture baseline demographics

a. Age b. Sex c. Race d. Lesion counts - total, inflammatory, non-inflammatory e. FDA score

4. Efficacy evaluation

a. 5 point IGA score b. Total lesional count c. No. of inflammatory lesions d. No. of non-inflammatory lesions e. Photography (+-) f. Scoring of the Cardiff Acne Disability Index.

5. Safety Evaluation

a. Score of itchiness b. Score of scaling c. Score of erythema d. Score of pain

6. Primary end points -

a. percentage reduction in lesion counts from week 0 to week 8 i. total lesion counts ii. total inflammatory counts iii. total non-inflammatory counts b. Proportion of subjects who had a IGA score of 0 or 1 by week 8 c. Time to 50% reduction of total lesion counts

7. Secondary end point

a. Improvement of the Cardiff Acne Disability Index

Povidone Iodine will be applied on the face by the patient using his own finger tips - onto his acne affected areas on the face.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with mild to moderate inflammatory acne - grade 2 to 3.
2. Patients must be at least 12 years of age
3. No gender preference - both male and female allowed
4. Subjects who provide signed and dated written voluntary informed consent

Exclusion Criteria:

1. Thyroid Dysfunction
2. Pregnancy, Breast feeding
3. History of hypersensitivity to iodine
4. History of renal impairment
5. Using OCPs
6. Using concurrent medications known to exacerbate acne
7. Nodulocystic acne or other severe variants
8. Had a facial procedure - chemical or laser peel or microdermabrasion 2 weeks before the study
9. No topical antiacne products 2 weeks prior to study commencement till its conclusion.
10. No systemic corticosteroids 4 weeks prior to study start
11. No systemic retinoids 3 months prior to study start
12. No concurrent use of tanning booths or sunbathing
13. Any condition in the judgement of the investigator that may place the person at unacceptable risk for participation
14. Any subject who participated in another clinical trial with 30 days of study entry,

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
5 point Acne Score | 2 months
  0 Clear, indicating no inflammatory or noninflammatory lesions
  1. Almost clear, rare noninflammatory lesions with no more than one papules/pustule;
  2. Mild, some noninflammatory lesions, no more than a few papules/pustules but no nodules
  3. Moderate, up to many noninflammatory lesions, may have some inflammatory lesions, but no more than one small nodule;
  4. Severe, up to many noninflammatory and inflammatory lesions, but no more than a few nodules.
Lesional Counts | 2 months
  b. Total lesional count c. No. of inflammatory lesions d. No. of non-inflammatory lesions
Effect on Quality of Life | 2 months
  Scoring of the Cardiff Acne Disability Index.
Safety | 2 months
  1. Score of itchiness
  2. Score of scaling
  3. Score of erythema
  4. Score of pain

CONTACTS AND LOCATIONS:
Overall Officials: Sam SY Yang, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore